CLINICAL TRIAL: NCT02482883
Title: Evaluation of the Efficacy of Transcutaneous Trigeminal Nerve Stimulation for Prevention of Cerebral Vasospasm and Its Consequences After Subarachnoid Haemorrhage Due to Ruptured Aneurysm: a Multicentre, Randomized, Double-blind Study
Brief Title: Evaluation of Transcutaneous Trigeminal Nerve Stimulation for Prevention of Cerebral Vasospasm After Subarachnoid Haemorrhage
Acronym: TRIVASOSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TRIVASOSTIM
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Subarachnoid Haemorrhage (SAH)
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active Transcutaneous Electrical Nerve Stimulation (Active Comparator): Arm A, treated by active stimulation of the trigeminovascular system after placement of the TENS device.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- sham Transcutaneous Electrical Nerve Stimulation (Sham Comparator): Arm B, treated by non-active (sham) stimulation after placement of the TENS device. This absence of stimulation corresponds to the standard of care currently received by patients hospitalized for SAH due to ruptured aneurysm.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — All patients will undergo placement of a facial transcutaneous electrical nervous stimulation (TENS) device, but device activation will be randomized [active stimulation vs non-active (placebo) stimulation], for an initial period of 10 days.

SUMMARY:
Subarachnoid haemorrhage (SAH) secondary to ruptured aneurysm represents 5 to 15% of all cases of stroke. The mortality rate of SAH is 40% and the risk of serious neurological sequelae among survivors is 10 to 20%.The causes of morbidity and mortality are mainly related to the initial damage induced by SAH and delayed cerebral ischaemia (DCI), which is generally secondary to cerebral vasospasm.

Cerebral vasospasm is one of the main factors of poor prognosis after SAH, as it is associated with a 1.5- to 3-fold increase in the mortality rate during the 2 weeks following SAH in these patients.

Despite a significant improvement in the time to management of this disease and the fact that the ruptured aneurysm is very often rapidly excluded by surgical or endovascular intervention, patients who survive the initial SAH remain at risk of severe complications over the following 2 weeks.

Vascular stenosis of an arterial segment, called cerebral vasospasm, is observed in more than 70 to 95% of cases on digital subtraction angiography between the 7th and 14th days after ruptured aneurysm. This angiographic vasospasm can be responsible for cerebral infarction in 52 to 81% of cases.

Despite 50 years of research, no clearly demonstrated effective treatment for vasospasm is currently available.

This is a multicentre, randomized, comparative study, including 364 patients during the acute phase following ruptured aneurysm, in whom management is very often limited to control of complications, after exclusion of the aneurysm.

The objective of this study is to validate the efficacy of transcutaneous trigeminal nerve stimulation for the prevention of vasospasm and limitation of the consequences of delayed cerebral ischaemia after SAH.

This is an innovative project, as it comprises intervention in these patients prior to the development of complications and could limit the development of these complications. The prevention tool, based on external facial nerve stimulation, is a totally innovative, reversible and noninvasive technique. Use of nerve stimulation in this indication has never been previously reported and could radically modify the intensive care management of this disease over the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* Admission within 48 h after onset of SAH.
* Ruptured cerebral aneurysm confirmed on CT angiography or cerebral angiography.
* Patient classified as grade I-IV according to the WFNS (World Federation of Neurological Surgeons) classification.
* Covered by French national health insurance.
* Absence of active cancer.

Exclusion Criteria:

* Age < 18 years and > 75 years.
* Absence of signature of the informed consent form by the patient or a close relative.
* Person subject to reinforced protection Clinical state on admission classified as WFNS grade V (excessively high mortality rate).
* Intracerebral or intraventricular haemorrhage without subarachnoid involvement.
* Major complication during the aneurysm exclusion procedure.
* SAH with no demonstrated aneurysm.
* Presence of non-ruptured cerebral aneurysm.
* Contraindication to placement of a transcutaneous device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Development of cerebral Infarction on MRI (FLAIR sequence) | At 3 months

SECONDARY OUTCOMES:
Functional disability (modified Rankin scale and GOS). | At 6 months
Evaluation of quality of life (EQ-5D) | At 6 months
An anomaly of perfusion detected on perfusion CT-scan | At day 6
Evaluation of MTT (Mean Transit Time) | At day 6

CONTACTS AND LOCATIONS:
Overall Officials: Benoit BATAILLE, Principal Investigator — Poitiers University Hospital
Locations (1):
- BATAILLE, Poitiers, France